CLINICAL TRIAL: NCT04274972
Title: The Microbiome of Pancreatic Cancer: "PANDEMIC" Study
Acronym: PANDEMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: 2480CESC
Record Dates: First submitted 2020-02-17; First posted 2020-02-18 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Microbial Colonization; Pancreas Cancer; Pancreas Infection; Pancreas; Fistula
MeSH Terms: conditions — Communicable Diseases; Pancreatic Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreaticoduodenectomy patients: All patients, affected by a resectable PDAC of the head of the pancreas, visited at the Department of Pancreatic Surgery of Verona, will be enrolled. All the patients must be scheduled for an elective PD. The oral and rectal microbiome samples will be collected preoperatively. The PDAC tissue from the surgical specimen, the intestinal mucosal tissue from the enteric side of the pancreatic anastomosis, and the bile sample will be collected intraoperatively. On the 30th postoperative day, the oral and rectal samples will be repeated.
  Interventions: Diagnostic Test: Microbiome evaluation

INTERVENTIONS:
Diagnostic Test: Microbiome evaluation — The oral and rectal microbiome samples will be collected preoperatively. The PDAC tissue from the surgical specimen, the intestinal mucosal tissue from the enteric side of the pancreatic anastomosis, and the bile sample will be collected intraoperatively. On the 30th postoperative day, the oral and rectal samples will be repeated

SUMMARY:
Microbiome in patients affected by pancreatic ductal adenocarcinoma may present specific and identifiable patterns. These variations could affect the surgical outcome and increase the risk of life-threatening infections supported by multidrug-resistant bacteria. The identification of microbial signatures with tumor specificity may have a potential role in postoperative risk stratification. Variation of pancreatic, intestinal or bile microbiome and their relationship can be investigated and measured as promising tools in order to predict and overcome the clinical and infectious burden imposed by MDR infections. The prospect of a potential role for probiotics to promote competition against the pathogens and to improve the gastrointestinal barrier integrity has also been raised. Moreover, if the bacterial composition in human PDAC was confirmed to be distinct from that of the normal pancreas, microbiome variation could be used as a potential biomarker, to assess the potential for malignancy in precursor neoplastic lesions. However, we believe that a preliminary and explorative study is necessary. The study aims to outline the pancreatic microbiome of patients who undergo upfront PD for resectable PDAC and to characterize the possible association between bacterial composition and the occurrence of post-operative complications, particularly POPF and IC.

DETAILED DESCRIPTION:
Pancreatic cancer is predicted to become the second leading cause of cancer-related death in the western world by 2030. Patients still have a poor prognosis, and a complete surgical resection provides the only potential for long-term cure of pancreatic ductal adenocarcinoma (PDAC) with a 5-year survival of only around 20%.

In addition, despite all the advances and technical modifications developed during this past decade, pancreatic surgery is still hampered by considerable postoperative morbidity. Postoperative pancreatic fistula (POPF), with a range of incidence between 3-45%, and the infectious complications (IC) that occur in nearly one-third of the patients are still the more frequent and dreadful complications after pancreatic resection. Moreover, in patients submitted to pancreaticoduodenectomy (PD), the constantly growing presence of multidrug-resistant (MDR) bacteria increases the morbidity and mortality rate. Those complications may also limit access to adjuvant chemotherapy and result in higher costs and longer hospitalization.

The high clinical burden of pancreatic surgery, associated with the overall poor outcome of PDAC and worldwide diffusion of antibiotic resistance, suggest the urgent need to enhance our knowledge on new and modifiable risk factors able to affect the surgical, the infectious and the oncological outcomes.

The alteration of the microbiome recently emerged as a contributor to oncogenesis, as a risk factor for postoperative morbidity in many intestinal tract malignancies and as one of the leading causes of colonization by resistant pathogenic bacteria. Recent evidence suggests that the pancreas also harbors its microbiome and in PDAC this is markedly more abundant and with different patterns compared to a normal pancreas in both mice and humans. However, the intestinal and PDAC microbiome have never been compared in humans. Alteration of the microbiome induces an adaptive immune suppression and promotes an inflammatory status. Growing literature evidence shows that the microbiome accounts for local and systemic microenvironment changes. These alterations, characterized by immune suppression and selection of potentially pathogenic bacteria, may lead both to adverse outcomes after surgical treatment and to the overgrowth of multidrug-resistant flora.

Nevertheless, the etiologic relationship between intrapancreatic microbiota and postoperative complications in PDAC patients subjected to surgery has not yet been described.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years;
* PDAC lesion of the pancreatic head confirmed by preoperative histology or cytology;
* Scheduled for elective PD;
* ASA score < 4
* The ability of the subject to understand the character and individual consequences of the clinical trial
* Written informed consent

Exclusion Criteria:

* Patients with a degenerated pancreatic cyst lesion
* Neoadjuvant treatment (both radio and chemotherapy)
* Other current malignancies
* Antibiotic therapy during 4 weeks before surgery
* History of gastrointestinal tract resections or chronic gastrointestinal diseases
* Pregnant or breastfeeding patients
* Patients undergoing emergency surgery
* ASA score > 4
* Impaired mental state or language problems

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients, affected by a resectable PDAC of the head of the pancreas, visited at the Department of Pancreatic Surgery of Verona, will be enrolled. All the patients must be scheduled for an elective PD. The patients will be submitted to the routinely diagnostic preoperative work-up.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome evaluation | 30th day after surgery
  Qualitative and quantitative analysis of the pancreatic microbiome in patients with PDAC submitted to pancreaticoduodenectomy, sampling intraoperatively the lesion

SECONDARY OUTCOMES:
Microbiome samples correlation | 30th day after surgery
  Definition of a correlation between the pancreatic microbiome and the oral, bile, and rectal microbiome samples
Microbiome correlation to surgical outcomes | 90th day after surgery
  Definition of a correlation between the pancreatic microbiome and the development of the postoperative complications, particularly pancreatic fistula and infectious complications
Microbiome long-term evaluation | 90th day after surgery
  Identification of potential change in the microbiome after surgical resection, comparing pre and post-surgical oral and rectal samples

CONTACTS AND LOCATIONS:
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided